CLINICAL TRIAL: NCT00067145
Title: Computer Intervention for Prevention of Weight Regain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: COMINTER (completed)
Record Dates: First submitted 2003-08-11; First posted 2003-08-13 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

INTERVENTIONS:
Behavioral: Face-to-face maintenance program
Behavioral: Internet maintenance program

SUMMARY:
Many overweight patients are able to lose weight successfully, but then regain their weight. The purpose of this study is to develop and test the efficacy of 2 interventions to prevent weight regain in individuals who have recently lost weight. The two interventions being tested are a face-to-face group maintenance program and an Internet intervention. These interventions will be compared to a no-contact control group that receives quarterly newsletters. The primary outcome measure is weight regain from baseline to 18-months.

ELIGIBILITY:
10% weight loss in past 2 years

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300

CONTACTS AND LOCATIONS:
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Result] Wing RR, Tate DF, Gorin AA, Raynor HA, Fava JL. A self-regulation program for maintenance of weight loss. N Engl J Med. 2006 Oct 12;355(15):1563-71. doi: 10.1056/NEJMoa061883. PMID 17035649
- [Derived] Marinilli Pinto A, Gorin AA, Raynor HA, Tate DF, Fava JL, Wing RR. Successful weight-loss maintenance in relation to method of weight loss. Obesity (Silver Spring). 2008 Nov;16(11):2456-61. doi: 10.1038/oby.2008.364. Epub 2008 Aug 14. PMID 18719680
- See also: Related Info — http://www.weightresearch.org